CLINICAL TRIAL: NCT02453919
Title: Register of Cardiovascular Complications Among People Living With HIV
Acronym: RECOVIH
Status: Recruiting | Type: Observational
Sponsor: Saint Antoine University Hospital (Other)
Responsible Party: Principal Investigator, Franck Boccara, MD, PhD, Saint Antoine University Hospital
Other Study IDs: RECOVIH
Record Dates: First submitted 2015-05-19; First posted 2015-05-27 (Estimated); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: HIV; Cardiovascular Diseases
Keywords: functional cardiac abnormality; morphologic cardiac abnormality; blood pressure abnormality
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RECOVIH: Complete cardiac examination including echocardiography, ischemia tests, and ambulatory blood pressure monitoring.
  Collection of clinical information and biochemical laboratory results.

SUMMARY:
The REgister of cardiovascular COmplications among people living with HIV (RECOVIH) is a single hospital registry of adults living with HIV, with one or more other cardiovascular risk factor, who undergo cardiac examination at the Cardiac Center of the Saint Antoine Hospital.

RECOVIH is an observational and prospective, monocentric (institutional) registry, with anonymized cardiac, biochemical and associated data collection.

DETAILED DESCRIPTION:
This hospital-based cardiac registry maintains data from all non-opposing adults living with HIV, with one or more other cardiac risk factor, who undergo complete cardiac examination at the Cardiac Center at the Saint Antoine Hospital.

RECOVIH registry:

The focus of this hospital-based cardiac registry is on clinical care, particularly on risk stratification, of adults living with HIV.

The register was designed to evaluate echocardiographic, coronarographic, and blood pressure abnormalities among people living with HIV (PLWH).

The primary goal of this single hospital registry is the improvement of patient care, especially risk stratification, by medical audit-type evaluation of cardiac tests and outcomes.

RECOVIH data and research:

Cardiac, biochemical, and associated data collected by this single hospital registry are also used as a source of data for some types of research. This research is particularly timely and relevant as currently little scientific evidence exists describing optimal cardiac care, and risk stratification, for adults living with HIV.

The primary goal of research using RECOVIH data is the quantification of morphologic and functional cardiac abnormalities and blood pressure abnormalities.

The secondary research goal is the identification and description of key aspects of the relationship between HIV, cardiovascular diseases (CVD), and CVD risk factors. Exploration of this complex relationship may help identify and describe the impact of chronic HIV related infection and inflammation, antiretroviral use (ARV), and individual health risks on the development and course of morphologic and functional cardiac abnormalities and blood pressure levels.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Known HIV-1 seropositivity for minimum of six months (confirmed by Elisa and Western Blot)
* Underwent complete cardiac examination (echocardiography, ischemia test, ambulatory blood pressure monitoring) between 2005 and 2010 at the Cardiac Center in the Saint Antoine University Hospital in Paris, France
* Presenting a minimum of two cardiovascular risk factors (HIV and a minimum of one other) according to the AFFSSAPS 2005 and Morlat Report 2013.
* Willing and able to give informed consent to participate in the study

Exclusion Criteria :

* Refusal to give or sign informed consent
* Not associated with a social security regime (no health insurance)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults living with HIV in Paris, France who have a minimum of one additional cardiovascular risk factor and underwent complete cardiac examination at the Cardiac Center of the Saint Antoine University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2010-02 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular mortality | 20 years
  Cardiovascular mortality as classified using the 10th revision of the International Classification of Diseases (cardiovascular diagnosis codes I 00-I 99).

SECONDARY OUTCOMES:
Echocardiographic profile (composite) | 20 years
  Parameters concerning - left ventricular dysfunction both systolic and diastolic, valvulopathies, pulmonary pressure, pericardial involvement under cross-sectional echocardiography and tissue Doppler imaging.
Ischemia profile (composite) | 20 years
  Parameters of ischemia tests including - exercise tolerance test, and stress-echocardiography under dobutamine or exercise.
Blood pressure profile (composite) | 20 years
  Parameters from - ambulatory blood pressure monitoring over 24 hours using a Pressure Holter.

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Cohen, MD, PhD, Study Chair — Saint Antoine University Hospital
Locations (1):
- Division of Cardiology, Saint Antoine University Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wever Pinzon O, Silva Enciso J, Romero J, Makani H, Fefer J, Gandhi V, Bangalore S, Chaudhry FA. Risk stratification and prognosis of human immunodeficiency virus-infected patients with known or suspected coronary artery disease referred for stress echocardiography. Circ Cardiovasc Imaging. 2011 Jul;4(4):363-70. doi: 10.1161/CIRCIMAGING.110.961060. Epub 2011 Jul 12. PMID 21750273
- [Background] Mariano-Goulart D, Jacquet JM, Molinari N, Bourdon A, Benkiran M, Sainmont M, Cornillet L, Macia JC, Reynes J, Ben Bouallegue F. Should HIV-infected patients be screened for silent myocardial ischaemia using gated myocardial perfusion SPECT? Eur J Nucl Med Mol Imaging. 2013 Jan;40(2):271-9. doi: 10.1007/s00259-012-2262-1. Epub 2012 Nov 14. PMID 23149821
- [Background] Duong M, Cottin Y, Piroth L, Fargeot A, Lhuiller I, Bobillier M, Grappin M, Buisson M, Zeller M, Chavanet P, Wolf JE, Portier H. Exercise stress testing for detection of silent myocardial ischemia in human immunodeficiency virus-infected patients receiving antiretroviral therapy. Clin Infect Dis. 2002 Feb 15;34(4):523-8. doi: 10.1086/338398. Epub 2002 Jan 2. PMID 11797181
- [Background] Catzin-Kuhlmann A, Orea-Tejeda A, Castillo-Martinez L, Colin-Ramirez E, Asz D, Aguirre VH, Herrera LE, Valles V, Aguilar-Salinas CA, Sierra J, Calva JJ. Human immunodeficiency virus-infected subjects have no altered myocardial perfusion. Int J Cardiol. 2007 Oct 31;122(1):90-2. doi: 10.1016/j.ijcard.2006.11.040. Epub 2007 Jan 26. PMID 17258826
- [Background] Mansoor A, Golub ET, Dehovitz J, Anastos K, Kaplan RC, Lazar JM. The association of HIV infection with left ventricular mass/hypertrophy. AIDS Res Hum Retroviruses. 2009 May;25(5):475-81. doi: 10.1089/aid.2008.0170. PMID 19397399
- [Background] Mondy KE, Gottdiener J, Overton ET, Henry K, Bush T, Conley L, Hammer J, Carpenter CC, Kojic E, Patel P, Brooks JT; SUN Study Investigators. High Prevalence of Echocardiographic Abnormalities among HIV-infected Persons in the Era of Highly Active Antiretroviral Therapy. Clin Infect Dis. 2011 Feb 1;52(3):378-86. doi: 10.1093/cid/ciq066. Epub 2010 Dec 9. PMID 21217185
- [Background] Reinsch N, Neuhaus K, Esser S, Potthoff A, Hower M, Brockmeyer NH, Erbel R, Neumann T; German Competence Network for Heart Failure; German Competence Network for HIV AIDS. Prevalence of cardiac diastolic dysfunction in HIV-infected patients: results of the HIV-HEART study. HIV Clin Trials. 2010 May-Jun;11(3):156-62. doi: 10.1310/hct1103-156. PMID 20739268
- [Background] Neumann T, Esser S, Potthoff A, Pankuweit S, Neumann A, Breuckmann F, Neuhaus K, Kondratieva J, Buck T, Muller-Tasch T, Wachter R, Prettin C, Gelbrich G, Herzog W, Pieske B, Rauchhaus M, Loffler M, Maisch B, Mugge A, Wasem J, Gerken G, Brockmeyer NH, Erbel R; HIV-HEART Study Investigative Group. Prevalence and natural history of heart failure in outpatient HIV-infected subjects: rationale and design of the HIV-HEART study. Eur J Med Res. 2007 Jun 27;12(6):243-8. PMID 17666313
- [Background] Reinsch N, Buhr C, Krings P, Kaelsch H, Kahlert P, Konorza T, Neumann T, Erbel R; Competence Network of Heart Failure. Effect of gender and highly active antiretroviral therapy on HIV-related pulmonary arterial hypertension: results of the HIV-HEART Study. HIV Med. 2008 Aug;9(7):550-6. doi: 10.1111/j.1468-1293.2008.00602.x. Epub 2008 Jun 28. PMID 18557952
- [Background] Martinez-Garcia T, Sobrino JM, Pujol E, Galvez J, Benitez E, Giron-Gonzalez JA. Ventricular mass and diastolic function in patients infected by the human immunodeficiency virus. Heart. 2000 Dec;84(6):620-4. doi: 10.1136/heart.84.6.620. PMID 11083740
- [Background] Hsue PY, Hunt PW, Ho JE, Farah HH, Schnell A, Hoh R, Martin JN, Deeks SG, Bolger AF. Impact of HIV infection on diastolic function and left ventricular mass. Circ Heart Fail. 2010 Jan;3(1):132-9. doi: 10.1161/CIRCHEARTFAILURE.109.854943. Epub 2009 Nov 20. PMID 19933410
- [Background] Oliviero U, Bonadies G, Bosso G, Foggia M, Apuzzi V, Cotugno M, Valvano A, Leonardi E, Borgia G, Castello G, Napoli R, Sacca L. Impaired diastolic function in naive untreated human immunodeficiency virus infected patients. World J Cardiol. 2010 Apr 26;2(4):98-103. doi: 10.4330/wjc.v2.i4.98. PMID 21160704
- [Background] Lewden C, May T, Rosenthal E, Burty C, Bonnet F, Costagliola D, Jougla E, Semaille C, Morlat P, Salmon D, Cacoub P, Chene G, Group AEMS, Mortavic. Changes in causes of death among adults infected by hiv between 2000 and 2005: The
- [Background] Palella FJ Jr, Baker RK, Moorman AC, Chmiel JS, Wood KC, Brooks JT, Holmberg SD; HIV Outpatient Study Investigators. Mortality in the highly active antiretroviral therapy era: changing causes of death and disease in the HIV outpatient study. J Acquir Immune Defic Syndr. 2006 Sep;43(1):27-34. doi: 10.1097/01.qai.0000233310.90484.16. PMID 16878047
- [Background] Dube MP, Stein JH, Aberg JA, Fichtenbaum CJ, Gerber JG, Tashima KT, Henry WK, Currier JS, Sprecher D, Glesby MJ; Adult AIDS Clinical Trials Group Cardiovascular Subcommittee; HIV Medical Association of the Infectious Disease Society of America. Guidelines for the evaluation and management of dyslipidemia in human immunodeficiency virus (HIV)-infected adults receiving antiretroviral therapy: recommendations of the HIV Medical Association of the Infectious Disease Society of America and the Adult AIDS Clinical Trials Group. Clin Infect Dis. 2003 Sep 1;37(5):613-27. doi: 10.1086/378131. Epub 2003 Aug 15. No abstract available. PMID 12942391
- [Background] Aberg JA, Gallant JE, Ghanem KG, Emmanuel P, Zingman BS, Horberg MA; Infectious Diseases Society of America. Primary care guidelines for the management of persons infected with HIV: 2013 update by the HIV medicine association of the Infectious Diseases Society of America. Clin Infect Dis. 2014 Jan;58(1):e1-34. doi: 10.1093/cid/cit665. Epub 2013 Nov 13. PMID 24235263
- [Background] Lundgren JD, Battegay M, Behrens G, De Wit S, Guaraldi G, Katlama C, Martinez E, Nair D, Powderly WG, Reiss P, Sutinen J, Vigano A; EACS Executive Committee. European AIDS Clinical Society (EACS) guidelines on the prevention and management of metabolic diseases in HIV. HIV Med. 2008 Feb;9(2):72-81. doi: 10.1111/j.1468-1293.2007.00534.x. PMID 18257770
- [Background] Prise en charge médical des personnes vivants avec le VIH. Recommandations du groupe d'experts. Sous la direction du Pr Philippe Morlat et sous l'égide du CNS et de l'ANRS. www.cns.sante.fr. 2013.
- [Background] European Association for Cardiovascular Prevention & Rehabilitation; Reiner Z, Catapano AL, De Backer G, Graham I, Taskinen MR, Wiklund O, Agewall S, Alegria E, Chapman MJ, Durrington P, Erdine S, Halcox J, Hobbs R, Kjekshus J, Filardi PP, Riccardi G, Storey RF, Wood D; ESC Committee for Practice Guidelines (CPG) 2008-2010 and 2010-2012 Committees. ESC/EAS Guidelines for the management of dyslipidaemias: the Task Force for the management of dyslipidaemias of the European Society of Cardiology (ESC) and the European Atherosclerosis Society (EAS). Eur Heart J. 2011 Jul;32(14):1769-818. doi: 10.1093/eurheartj/ehr158. Epub 2011 Jun 28. PMID 21712404
- [Background] Nayak G, Ferguson M, Tribble DR, Porter CK, Rapena R, Marchicelli M, Decker CF. Cardiac diastolic dysfunction is prevalent in HIV-infected patients. AIDS Patient Care STDS. 2009 Apr;23(4):231-8. doi: 10.1089/apc.2008.0142. PMID 19281430
- [Background] El Hattaoui M, Charei N, Boumzebra D, Aajly L, Fadouach S. [Prevalence of cardiomyopathy in HIV infection: prospective study on 158 HIV patients]. Med Mal Infect. 2008 Jul;38(7):387-91. doi: 10.1016/j.medmal.2008.03.006. Epub 2008 Jun 25. French. PMID 18583077
- [Background] Karavidas A, Foukarakis M, Lazaros G, Chini M, Fotiadis I, Arapi S, Gialernios T, Potamitis N, Gargalianos P, Matsakas E, Stefanadis C. Assessment of cardiac function with Doppler tissue imaging in asymptomatic HIV-infected patients. Int J STD AIDS. 2008 Apr;19(4):227-31. doi: 10.1258/ijsa.2007.007225. PMID 18482939
- [Background] Thoni GJ, Schuster I, Walther G, Nottin S, Vinet A, Boccara F, Mauboussin JM, Rouanet I, Ederhy S, Dauzat M, Messner-Pellenc P, Obert P. Silent cardiac dysfunction and exercise intolerance in HIV+ men receiving combined antiretroviral therapies. AIDS. 2008 Nov 30;22(18):2537-40. doi: 10.1097/QAD.0b013e328319806d. PMID 19005278
- [Background] Lang S, Mary-Krause M, Cotte L, Gilquin J, Partisani M, Simon A, Boccara F, Costagliola D; Clinical Epidemiology Group of the French Hospital Database on HIV. Impact of individual antiretroviral drugs on the risk of myocardial infarction in human immunodeficiency virus-infected patients: a case-control study nested within the French Hospital Database on HIV ANRS cohort CO4. Arch Intern Med. 2010 Jul 26;170(14):1228-38. doi: 10.1001/archinternmed.2010.197. PMID 20660842
- [Background] Fihn SD, Gardin JM, Abrams J, Berra K, Blankenship JC, Dallas AP, Douglas PS, Foody JM, Gerber TC, Hinderliter AL, King SB 3rd, Kligfield PD, Krumholz HM, Kwong RY, Lim MJ, Linderbaum JA, Mack MJ, Munger MA, Prager RL, Sabik JF, Shaw LJ, Sikkema JD, Smith CR Jr, Smith SC Jr, Spertus JA, Williams SV; American College of Cardiology Foundation; American Heart Association Task Force on Practice Guidelines; American College of Physicians; American Association for Thoracic Surgery; Preventive Cardiovascular Nurses Association; Society for Cardiovascular Angiography and Interventions; Society of Thoracic Surgeons. 2012 ACCF/AHA/ACP/AATS/PCNA/SCAI/STS Guideline for the diagnosis and management of patients with stable ischemic heart disease: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines, and the American College of Physicians, American Association for Thoracic Surgery, Preventive Cardiovascular Nurses Association, Society for Cardiovascular Angiography and Interventions, and Society of Thoracic Surgeons. J Am Coll Cardiol. 2012 Dec 18;60(24):e44-e164. doi: 10.1016/j.jacc.2012.07.013. Epub 2012 Nov 19. No abstract available. PMID 23182125
- [Background] Arbab-Zadeh A. Stress testing and non-invasive coronary angiography in patients with suspected coronary artery disease: time for a new paradigm. Heart Int. 2012 Feb 3;7(1):e2. doi: 10.4081/hi.2012.e2. Epub 2012 Feb 8. PMID 22690295